CLINICAL TRIAL: NCT04302948
Title: Rapid HCV RNA Testing and LInkage to Care
Acronym: TEAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 quarantines disrupted study and funding ended.
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Kimberly Page, Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-232
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Diagnostics; Point-of-care system
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Study staff who abstract outcomes from medical record will not be aware of patients' study arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): TaU includes screening for anti-HCV using a rapid point-of-care (PoC) test to screen for exposure to HCV followed by counseling, brief education and referral to provider for further evaluation for HCV treatment.
- Rapid PoC RNA testing (Experimental): Intervention arm includes Tau ( screening for anti-HCV using a rapid point-of-care (PoC) test, and a rapid PoC screening test for HCV RNA, counseling plus, brief education and referral to a provider for further evaluation for HCV treatment. Rapid HCV RNA testing will be conducted using Cepheid Xpert (r) system.
  Interventions: Other: HCV RNA screening

INTERVENTIONS:
Other: HCV RNA screening — The Cepheid Xpert testing requires a fingerstick to obtain blood spots which are then tested for HCV RNA. Results available within one to two hours, facilitating counseling for patients to link to care.
  Other Names: Cepheid Xpert system
  Arms: Rapid PoC RNA testing

SUMMARY:
The investigators propose to conduct a pilot randomized controlled trial comparing treatment as usual (TaU) for HCV screening (rapid anti-HCV screening and referral) to a intervention screening that includes TaU plus a rapid point-of-care HCV RNA test in persons experiencing homelessness. The primary outcome of interest is linkage-to-care. Linkage to care is defined as evaluation by a health care provider for HCV infection within 30 days of baseline screening and referral. We will compare the proportion of patients who are evaluated by a provider within the 30 day window in each study arm: (1) participants who screened positive with rapid anti-HCV and are referred for evaluation) and (2) Rapid HCV RNA plus TaU (those who tested positive with both rapid anti-HCV and confirmatory RNA and are also referred to a provider.) Secondarily, the investigators will also assess HCV RNA levels in both groups twelve weeks after treatment ends (24 to 36 weeks after anti-HCV screening) to determine the percent of individuals who achieved sustained virologic response (SVR12), which is a marker for cure.

DETAILED DESCRIPTION:
* The goal of this study is to simplify the HCV testing process using combined rapid screening and confirmation in order to reduce early barriers and improve linkage to care among a vulnerable high-risk homeless population. The investigators are partnering with Albuquerque Health Care for the Homeless (AHCH) to conduct rapid testing and provide counseling, test results, and referrals directly on site.
* After Rapid HCV testing the investigators will randomize participants to 1) counseling and referral to a provider, or 2) Rapid RNA testing plus counseling and referrals to a provider.

The study's primary is to to assess linkage to care, which is the percent of subjects who are evaluated by a provider specifically for HCV infection in both groups. Linkage to care will be determined via medical chart abstraction 30 days after testing. The investigators hypothesize that there will be a 30% absolute difference in linkage to care between study arms, with a higher percent of participants in the combined rapid testing group being linked to a provider for evaluation relative to the control group (rapid anti-HCV alone).

* The study's second aim is exploratory in nature and sequentially follows the first aim. The investigators will also assess HCV Cascade of care in both group, and by medical chart abstraction (up to 36 weeks after study entry) to determine the number and proportion of individuals who achieved sustained virologic response (SVR12), which is a marker for cure.
* The study's third aim is a qualitative inquiry into the use of supportive services by participants during treatment. Such services may include social work, case management, patient navigation, participation in support groups, etc. The investigators will review medical charts for this information. The investigators are interested to see if more individuals in one study arm will access one or more of these supportive services compared to the other study arm.

ELIGIBILITY:
Inclusion Criteria:

- Report being homeless and meet the Albuquerque Healthcare for the homeless HCH operating definition of homeless

Exclusion Criteria:

* having stable housing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants in each study arm who are evaluated by a provider specifically for HCV infection after screening | Within 30 days of anti-HCV screening
  Evaluation HCV infection by a health care provider will be assessed as having attended a clinic visit based on medical record review

SECONDARY OUTCOMES:
The proportion of patients in each study arm who achieve sustained viral response (SVR-12) | 12 weeks after end of treatment, representative of 24-36 weeks after anti-HCV screening
  SVR-12 weeks after end of treatment based on medical record review.

OTHER OUTCOMES:
Proportion of patients in each study arm who have receive any HCV-treatment related support services | 24 to 36 weeks after anti-HCV screening
  Case-management, patient navigation, participation in support groups or other supportive services.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Albuquerque HealthCare for the Homeless, Albuquerque, New Mexico
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No